CLINICAL TRIAL: NCT06643390
Title: A Multiple Ascending Dose Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MK-2225 in Healthy Participants
Brief Title: A Study of MK-2225 in Healthy Participants (MK-2225-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2225-003; MK-2225-003 (Other: MSD)
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MK-2225 Panel A (Experimental): Participants receive MK-2225 Dose 1 subcutaneously (SQ) once every 2 weeks (Q2W) over the course of 8 weeks.
  Interventions: Drug: MK-2225
- MK-2225 Panel B (Experimental): Participants receive MK-2225 Dose 2 SQ Q2W over the course of 8 weeks based on the safety and tolerability of the previous starting dose.
  Interventions: Drug: MK-2225
- MK-2225 Panel C (Experimental): Participants receive MK-2225 Dose 3 SQ Q2W over the course of 8 weeks based on the safety and tolerability of the previous starting dose.
  Interventions: Drug: MK-2225
- MK-2225 Panel D (Experimental): Participants receive MK-2225 Dose 4 SQ Q2W over the course of 8 weeks based on the safety and tolerability of the previous starting dose.
  Interventions: Drug: MK-2225
- Placebo (Placebo Comparator): Participants receive placebo SQ Q2W over the MK-2225-matched time period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MK-2225 — Subcutaneous administration
  Arms: MK-2225 Panel A; MK-2225 Panel B; MK-2225 Panel C; MK-2225 Panel D
Other: Placebo — Subcutaneous administration
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn about the safety of MK-2225, including how well people tolerate it. Researchers also want to learn what happens to different doses of MK-2225 in a person's body over time.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Body Mass Index (BMI) ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* History of hypersensitivity to the MK-2225 drug substance, its inactive ingredients or the placebo (normal saline)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 20 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study/study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of MK-2225 | At designated timepoints (up to approximately 16 weeks)
  Blood samples will be collected to determine the Cmax of MK-2225.
Lowest Plasma Concentration (Ctrough) of MK-2225 | At designated timepoints (up to approximately 16 weeks)
  Blood samples will be collected to determine the Ctrough of MK-2225.
Time to Maximum Plasma Concentration (Tmax) of MK-2225 | At designated timepoints (up to approximately 16 weeks)
  Blood samples will be collected to determine the Tmax of MK-2225.
Area Under the Concentration-Time Curve from Time 0 to Tau (AUC0-τ) of MK-2225 | At designated timepoints (up to 16 approximately weeks)
  Blood samples will be collected to determine the AUC0-τ of MK-2225.
Apparent Terminal Half-life (t1/2) of MK-2225 | At designated timepoints (up to approximately 16 weeks)
  Blood samples will be collected to determine the t1/2 of MK-2225.
Mean Accumulation Ratio of MK-2225 | At designated timepoints (up to approximately 16 weeks)
  Blood samples will be collected at designated timepoints to determine the mean accumulation ratio of MK-2225.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami (Site 0002), Miami, Florida
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO (Site 0004), Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com